CLINICAL TRIAL: NCT02646969
Title: Growth and Metabolic Biomarkers of Healthy Term Infants Fed Formulas With Staged Protein Concentrations Over the First Year of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13.13.INF
Record Dates: First submitted 2015-11-06; First posted 2016-01-06 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2023-01

CONDITIONS: Healthy Term Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Formula regimen 1 (Active Comparator): Product Control from enrollment to transition phase 1 (blinded administration), followed by open label administration for 2 months.
  Product Test 2 from transition phase 2 to 1 year old (open label) Commercial follow up formula from 1 year old
  Interventions: Dietary Supplement: Formula regimen 1
- Formula regimen 2 (Active Comparator): Product Test 1 from enrollment to transition phase 1 (blinded administration) Product Control for 2 months(open label) Product Test 2 from transition phase 2 to 1 year old (open label) Commercial follow up formula from 1 year old
  Interventions: Dietary Supplement: Formula regimen 2
- Reference group (No Intervention): Infants fed HM exclusively through at least 4 months of age. Once breastfeeding is over and if wished Infant will receive Product test 2 until 1 year old followed by the commercial follow-up formula

INTERVENTIONS:
Dietary Supplement: Formula regimen 1
  Arms: Formula regimen 1
Dietary Supplement: Formula regimen 2
  Arms: Formula regimen 2

SUMMARY:
Growth and metabolic biomarkers of healthy term infants fed formulas with staged protein concentrations over the first year of life

DETAILED DESCRIPTION:
The overall objective of this study is to assess growth and biomarkers of energy and protein metabolism in healthy term infants fed with two different study formula regimens from birth to 12 months of age and to follow up the infants to 4 years of age.

ELIGIBILITY:
Inclusion Criteria:

Healthy infants will be enrolled in the study provided they meet the following inclusion criteria:

1. Having obtained his/her parents' (or his/her legally accepted representative's [LAR's]) written informed consent and having evidence of personally signed and dated informed consent document indicating that the infant's parents/LAR have been informed of all pertinent aspects of the study.
2. Age ≤ 7 days after birth (date of birth = Day 0)
3. Full-term gestational birth (≥ 37 and ≤ 42 weeks)
4. Born to mothers with pre-pregnancy body mass index (BMI) ≥ 18.5 and < 26 kg/m2
5. Born to mothers who independently elected, before study enrollment, not to breastfeed (not applicable for infants in the HM-fed comparator group)
6. Weight ≥ 2'500 g and ≤ 4'200 g
7. Infant's parent(s)/LAR is of legal age of consent, has sufficient command of French language to complete the informed consent and other study documents, and is willing and able to fulfill the requirements of the study protocol
8. Infant's parent(s)/LAR is able to be contacted directly by telephone throughout the study

Exclusion Criteria:

Infants who exhibit one or more of the following criteria are excluded from enrollment in the study:

1. Born to mothers with hormonal or metabolic disease (e.g. Type-1, Type-2, or gestational diabetes diagnosed according to standardized criteria)
2. Born to mothers who smoked > 10 cigarettes per day during pregnancy
3. Born to mothers who used illicit drugs (e.g. marijuana, cocaine, amphetamines, or heroin) or alcohol (> 3 alcoholic beverages per week) during pregnancy
4. Cognitive or physical developmental disorders (e.g. malabsorptive disorders such as short bowel syndrome; neurological and congenital disorders that may delay growth such as cerebral palsy, agenesis of the corpus callosum, spina bifida, Down Syndrome, Cri Du Chat; disorders that may lead to obesity such as Prader willi syndrome, Angelman syndrome; other renal, hepatic, pancreatic, or cardiovascular disorders)
5. Received radiation therapy (eg. scannography or interventional radiology)
6. Participation in any other clinical trial prior to enrollment
7. Infants or infant's family who in the Investigator's judgment cannot be expected to comply with the protocol or study procedures

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 691 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Growth velocity of formula regimen 1 and 2 versus WHO growth curve | 0-6 months
  Compare weight gain velocity (g/day) of each formula-fed group from enrollment to 6 months of age and compare to the World Health Organization (WHO) standards
Growth velocity (g/day) of formula regimen 1 and 2 versus a human milk (HM)-fed comparator group | 0-6 months
  Assess the growth velocity of each formula-fed group from enrollment to 6 months of age and compare to growth velocity of a human milk (HM)-fed comparator group.

SECONDARY OUTCOMES:
Growth velocity of formula regimen 1 and 2 versus WHO growth curve and versus a human milk (HM)-fed comparator group | 0-3 months and 0-12 months
  Assess the growth velocity of each formula-fed group from enrollment to 3 months, and from enrollment to 12 months, and compare to both WHO standards and to the HM-fed comparator group.
Other growth parameters z-scores of formula regimen 1 and 2 versus WHO standards and versus a human milk (HM)-fed comparator group | 6 and 12 months
  Weight-for-length, weight-for-age, length-for-age, head circumference-for-age, and BMI-for-age z-scores
Compare metabolic biomarkers measures in each formula-fed group to the HM-fed group | 0-4 years
  Assess and compare metabolic biomarkers in each formula-fed group to the HM-fed group. Here is the list of metabolic biomarkers that will be measured: free and total IGF-1, IGF-binding protein 2, IGF-binding protein 3, C-peptide, insulin, glucose, leptin, adiponectin, ghrelin in all subjects and complete amino acid profile in subset
Assess the adverse events (AEs) among all study subjects | 0-4 years
  Assess the type, incidence, severity, seriousness, and relationship to study formulas of AEs among study subjects.
Assess and compare the child behavior in each group until 4 years of age | 0-4 years
  Neurodevelopment will be assessed by parental ratings of child development using validated measures Ages and Stages Questionnaire (ASQ)
Assess and compare the neurodevelopment in each group until 4 years of age | 0-4 years
  Neurodevelopment will be assessed by tests of child development using validated Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV)
Body Composition: Body density [kg/L] using PeaPod | 1-6 months
  Body density in kg/L will be assessed using PeaPod
Body Composition: Body mass [kg] using PeaPod | 1-6 months
  Body mass in kg will be assessed using PeaPod
Body Composition: Body surface area [cm²] using PeaPod | 1-6 months
  Body surface area in cm² will be assessed using PeaPod
Body Composition: Body volume [L] using PeaPod | 1-6 months
  Body volume in L will be assessed using PeaPod
Body Composition: Fat free mass [kg] using PeaPod | 1-6 months
  Fat free mass in kg will be assessed using PeaPod
Body Composition: Fat free mass density [kg/L] using PeaPod | 1-6 months
  Fat free mass density in kg/L will be assessed using PeaPod
Body Composition: Fat mass [kg] using PeaPod | 1-6 months
  Fat mass in kg will be assessed using PeaPod
Body Composition: Percentage fat free mass using PeaPod | 1-6 months
  Percentage fat free mass will be assessed using PeaPod
Body Composition: Percentage fat mass using PeaPod | 1-6 months
  Percentage fat mass will be assessed using PeaPod
Body Composition: Thoracic gas volume (L) using PeaPod | 1-6 months
  Thoracic gas volume in L will be assessed using PeaPod
Body Composition: Bone area [cm²] using DEXA | 0-3 years
  Bone area in cm² will be assessed using DEXA
Body Composition: Bone Mineral Content [g] using DEXA | 0-3 years
  Bone Mineral Content in g will be assessed using DEXA
Body Composition: Bone Mineral Density [g/cm²] using DEXA | 0-3 years
  Bone Mineral Density in g/cm² will be assessed using DEXA
Body Composition: Fat Free Mass [g] using DEXA | 0-3 years
  Fat Free Mass in g will be assessed using DEXA
Body Composition: Fat mass [g] using DEXA | 0-3 years
  Fat mass in g will be assessed using DEXA
Body Composition: Lean mass [g] using DEXA | 0-3 years
  Lean mass in g will be assessed using DEXA
Body Composition: Percentage fat using DEXA | 0-3 years
  Percentage fat will be assessed using DEXA
Body Composition: Total mass [g] using DEXA | 0-3 years
  Total mass in g will be assessed using DEXA
Stool microbiota profile, and metabolomics endpoints in each group. Associations between microbiota and metabolomics profiles (serum, urine, and stool). | 0-4 years
  Stool microbiota profile (including proportion of fecal bifidobacteria and other bacterial species that may influence energy homeostasis), and metabolomics profile (metabolite sets related to energy recovery and protein and lipid metabolism assessed in blood, urine, and stool samples) in a subset.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Paoli, MSc, Study Chair — Nestlé Research
Locations (9):
- France (9):
  - CHU Pellegrin, Bordeaux, Bordeaux
  - Hospices Civils de LYON - Hôpital Femme Mère Enfant de Bron, Bron
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hospices Civils de LYON - Hopital de La Croix Rousse, Lyon
  - Assistance Publique-Hôpitaux de Marseille, Hôpital de la Conception, Marseille
  - Assistance Publique-Hôpitaux de Marseille, Hôpital NORD, Marseille
  - Centre Hospitalier du Belvédère, Mont-Saint-Aignan
  - CHU de Nancy - Hôpital Brabois, Nancy
  - CHU - Hôpitaux de ROUEN, Rouen

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831